CLINICAL TRIAL: NCT05019846
Title: Stereotactic Prostate Radiotherapy With or Without Androgen Deprivation Therapy, a Phase III, Multi-institutional Randomized-controlled Trial. The SPA Trial.
Brief Title: SRT Versus SRT+ADT in Prostate Cancer
Acronym: SPA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Marco Lorenzo Bonu (Other)
Collaborators: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Sponsor-Investigator, Marco Lorenzo Bonu, MD, Scientific coordinator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Organization: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPA Trial vers. 1.1; 2020-005754-23 (EudraCT Number)
Record Dates: First submitted 2021-08-02; First posted 2021-08-25 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
Keywords: SRT; ADT; SBRT; high risk prostate cancer; unfavourable intermediate risk prostate cancer; randomized trial
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SRT+ADT (Experimental): Patients in ARM A will be treated with SRT on the prostate (consecutive days or at alternate days to a total dose of 36.25 Gy administered in 5 fraction (7.25 Gy/fraction) + LHRH analogue (Triptoreline 22.5 mg). An anti-androgen drug (es. Bicalutamide 50 mg) must be administered daily starting from 7 days before LHRH analogue administration to 10 days after to prevent the flare effect
  Interventions: Drug: Triptorelin Embonate; Drug: Bicalutamide 50 mg
- SRT alone (No Intervention): Patients in ARM B will be treated with SRT on prostate alone at a total dose of 36.25 Gy administered daily or on alternate days in 5 fraction (7.25 Gy/fraction).

INTERVENTIONS:
Drug: Triptorelin Embonate — single administration before SRT starting
  Arms: SRT+ADT
Drug: Bicalutamide 50 mg — 1 dose each day, 7 days before LHRH until 10 days after LHRH administration
  Arms: SRT+ADT

SUMMARY:
To clarify the role of short-term Androgen deprivation therapy (ADT) in the context of intermediate unfavorable and a subclass of high-risk patients treated with prostate Stereotactic radiotherapy (SRT).

In intermediate unfavorable risk group, when choosing standard external beam radiotherapy, short term ADT is superior in terms of biochemical disease free survival (bDFS) to EBRT alone. In high risk disease, results of the combination therapy are even more clear. Prostate SRT has been endorsed as option for primary radical treatment for prostate cancer. In such patients, the benefit of ADT is still unknown and the decision is left to clinical judgement.

For these reasons, it seems to be relevant to propose a randomized, open label, phase III clinical trial of prostate SBRT + 6 months ADT versus prostate SBRT alone in intermediate unfavorable and a subgroup of high risk prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of prostate acinar adenocarcinoma with a minimum of 10 biopsy cores taken
* Prostate protocol MRI for local staging
* Patients belonging to intermediate unfavorable group according to the D'Amico/NCCN risk group classification:

  * -Grade group 3 or/and
  * -2-3 risk factors for intermediate category (PSA 10-20 ng/ml/ Grade group 2-3/ cT2b cT2c) or/and
  * -biopsy cores positive ≥50%
* Patients belonging to a subclass of high risk group according to the D'Amico/NCCN risk group classification:

  * -ISUP group 4 (GS 4+4, 3+5, 5+3) or
  * -cT3a stage or
  * PSA>20
* Eastern Coooperative Oncology Group (ECOG) PS 0-2
* Ability of the patient to understand and sign a written informed consent document
* Ability and willingness to comply with patients reported outcome questionnaires schedule during the study time
* IPSS 0-15
* Prostate Volume less than 100cc
* PSA must be dosed maximum 60 days before randomization
* No pathologic lymph nodes and distant metastasis on PET (fluorocholine) scan or CT scan+bone scan.
* Contraceptive measures for patients with partners with reproductive potential must be explained

Exclusion Criteria:

* History of Malignant tumors in the previous 2 years excluding non melanoma cancers of the skin. If a patient presents an anamnesis of malignancy (excluding non melanoma skin cancers) it must be free from disease since 24 months at the time of enrollement.
* Previous prostate surgery other than TURP (at least 6 weeks prior to start of SBRT).
* Previous pelvic RT
* Prior androgen deprivation therapy (excluding 5alpha reductase inhibitors)
* Any prior active treatment for prostate cancer; patients on previous active surveillance are eligible if inclusion criteria are met
* Active severe inflammatory bowel disease
* Bilateral hip prothesis or any implant that could seriously interfere with dosimetric calculations
* Age >80 years.
* cT4a, cT3b or pelvic lymph node involvement
* Controindication or hypersensitivity to the use of Triptoreline
* 5alpha reductase inhibitors not discontinued 4 weeks prior to randomization
* History of bone fractures and fall
* Risk factors for abnormal heart rhythms or QT prolongation.
* Use of concomitant medications that prolong the QT/QTc interval

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate cancer patients
Enrollment: 310 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
biochemical disease free survival | outcome will be evaluated at the completion of 5 years of follow-up
  form the date of the end of radiotherapy to the date of PSA meeting protocol criteria for biochemical relapse or last Follow-up visit. Outcome is mesured in months.

SECONDARY OUTCOMES:
Disease free survival | outcome will be evaluated at the completion of 5 years of follow-up
  from the date of the end of radiotherapy to the date of relapse (any) or last Follow-up visit.Outcome is mesured in months.
freedom from local recurrence | outcome will be evaluated at the completion of 5 years of follow-up
  from the date of the end of radiotherapy to the date of local relapse or last Follow-up visit. Outcome is mesured in months.
freedom from regional recurrence | outcome will be evaluated at the completion of 5 years of follow-up
  from the date of the end of radiotherapy to the date of regional relapse or last Follow-up visit. Outcome is mesured in months.
freedom from distant metastasis | outcome will be evaluated at the completion of 5 years of follow-up
  from the date of the end of radiotherapy to the date of metastatic relapse or last Follow-up visit. Outcome is mesured in months.
Overall survival | outcome will be evaluated at the completion of 5 years of follow-up
  from the date of the end of radiotherapy to the date of death 8any cause) or last Follow-up visit. Outcome is mesured in months.
quality of life, prostate related quality of life in prostate cancer | 12 weeks after SRT, 3, 6 and 12 months after SRT
  scored with questionnaire Expandend Prostate cancer Index Composite-26 (EPIC-26), score scale is 0-100 with higher scores representing better health related quality of life
quality of life, prostate related quality of life questionnarire | 12 weeks after SRT, 3, 6 and 12 months after SRT
  scored with questionnaire European organization for research and treatment of cancer PR 25, (EORTC PR 25), All of the scales and single-item measures range in score from 0 to 100. A high score for the Sexual Activity and Sexual Functioning scales represents a high level of functioning, whereas a high score for the Urinary, Bowel, and Hormonal Treatment Related symptoms scales and Incontinence Aid item represents a high level of symptomatology or problems.
patients reported outcome, erectile function assessment, | 12 weeks after SRT, 3, 6 and 12 months after SRT
  scored with questionnaire International Index of Erectile Function 5 (IIEF from 25 (best) to 5 (worse))
patients reported outcome, prostate related symptoms assessment | 12 weeks after SRT, 3, 6 and 12 months after SRT
  scored with questionnaire Internation Prostate syntoms scale (IPSS, from 0 (best) to 35 (worse))
Clinician reported Acute Toxicity, assessed with CTCAE 5.0 scales | from the beginning of treatment until 6 months after SRT
  Outcome is mesured in 0-5 scale (higher scale worse toxicity)
Clinician reported Late Toxicity, assessed with CTCAE 5.0 scales | from 6 months after SRT 5 years of follow-up
  Outcome is mesured in 0-5 scale (higher scale worse toxicity)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Triggiani, MD PHD, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- ASST Spedali Civili of Brescia, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: Yes
Concurrently with the publication of study results concerning efficacy, we will deliver a completely deidentified data set to an appropriate data archive for sharing purposes.
Supporting Information: Study Protocol
Time Frame: Concurrently with the publication of study results concerning efficacy, we will deliver a completely deidentified data set to an appropriate data archive for sharing purposes.
Access Criteria: explicit request
URL: http://dm.radioterapiabs@gmail.com